CLINICAL TRIAL: NCT05935319
Title: The Effectiveness of a VIVIFRAIL Program in Improving the Frailty and Physical Function in the Elderly
Brief Title: VIVIFRAIL Program in Improving the Frailty and Physical Function in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, WangJiaJie, Principal Investigator, Mennonite Christian Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Huang Xin-en
Record Dates: First submitted 2023-06-07; First posted 2023-07-07 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2024-07

CONDITIONS: Frailty; Physical Activity; Cognitive Function
MeSH Terms: conditions — Frailty; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- experimental group (Experimental): Vivifrail
  Interventions: Other: Vivifrail
- control group (No Intervention): Traditional Sports Health Leaflet

INTERVENTIONS:
Other: Vivifrail — Assess the physical activity status of the elderly, use the Vivifrail grade, provide exercise intervention, and improve physical activity function.
  Arms: experimental group

SUMMARY:
The global population is aging, and Taiwan has become an aging society. The aging population continues to rise. When the physical function and mental state of the elderly gradually decline, it is easy for the elderly to enter a state of physical weakness. Weakness is the decline in the reserve capacity of the physiological system. It is also related to geriatric syndrome, causing falls, hospitalization, disability, death, and increased medical costs, burden on primary caregivers, and reduced quality of life for the elderly.

Physical exercise training has been considered to be an effective strategy to prevent and delay disability and frailty, so this study uses the Vivifrail program for the elderly. A family-based 12-week exercise program, including: resistance, strength, balance, flexibility and cardiorespiratory endurance exercise training, performed five days a week, at least 45-60 minutes each time, so that the elderly can exercise at home, It can also improve physical function and improve the quality of life.

This study adopts a randomized controlled trial (RCT) with a one-group pretest-posttest design, with pre-frail and frail elderly as the research objects, and uses comprehensive assessment of the elderly to understand the physical function of the elderly Status, Vivifrail for the elderly was provided for abnormal physical function items, and post-test evaluation was carried out 4 weeks and 12 weeks after the intervention. In Taiwan, there is no research on Vivifrail for the frail elderly. In view of this, it is hoped that through the Vivifrail program and the follow-up of case managers, multi-faceted and continuous integrated care can be provided. Improve and maintain the physical function of the frail elderly for reference in the daily care of the elderly in the future.

ELIGIBILITY:
Inclusion Criteria:

1. ≧65 years old and above.
2. Pre-frail and frail cases assessed by Frail Fried's frail phenotype.
3. Clear consciousness, willing to accept interviewers, able to communicate in Chinese and Taiwanese.
4. Those who can cooperate with physical activities and have ADL ≥ 60 points.

Exclusion Criteria:

1. Those who cannot cooperate with the interventional care plan.
2. Elderly who are seriously ill or terminally ill.
3. People living in institutions.
4. Incompatibility and exclusion: acute myocardial infarction or recent unstable angina, poorly controlled atrial or ventricular arrhythmia, dissected aortic aneurysm, severe aortic stenosis, endocarditis/acute cardiac Capsulitis, uncontrolled hypertension, acute thromboembolism, acute or severe heart failure, acute or severe respiratory failure, uncontrolled postural hypotension, acute incompensated diabetes mellitus, or uncontrolled hypoglycemia, past month There is a fracture (muscle strength training).

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 200 (Actual)
Dates: Start 2023-05-26 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Hand Grip | 1-2 minutes
  Grip strength defined as <28 kg for men and <18 kg for women
Short Physical Performance Battery(SPPB) | 5-10 minutes
  ≦9 points abnormal, 10-12 normal.
Activities of Daily Living(ADL) | 2-5 minutes
  The full score is 100 points, 0-20 points are completely dependent, 21-60 points are heavily dependent, 61-90 points are moderately dependent, 91-99 points are slightly dependent, and 100 points are completely independent.
Instrumental Activities of Daily Living(IADL) | 2-5 minutes
  The full score is 8 points, the higher the score, the better the function.
Mini-Mental State Examination(MMSE) | 10-20 minutes
  junior high school ≧ 24 points, elementary school ≧ 21 points, those without education ≧ 16 points.
Geriatric Depression Scale(GDS- 15) | 10-20 minutes
  The full score is 15 points, 0-4 points are normal, 5-9 points are mild depression, 10-14 points are moderate depression, and more than 15 points are depression.

CONTACTS AND LOCATIONS:
Overall Officials: Xin-en Huang, Principal Investigator — Host
Locations (1):
- WangJiaJie, Hualien City, Taiwan

IPD SHARING:
Plan to Share IPD: No